CLINICAL TRIAL: NCT06922435
Title: Evaluation of Management and Outcomes of Normal Labor in Eldakhla Hospital.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Abdel Baset Ahmed, Residant doctor, Assiut University
Other Study IDs: M &O normal labor Eldakhla
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Normal Labour

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group A: Patients with full-term labour

SUMMARY:
Labour is a physiologic process during which the products of conception are expelled outside of the uterus. Labour is achieved with changes in the biochemical connective tissue and with gradual effacement and dilatation of the uterine cervix as a result of rhythmic uterine contractions of sufficient frequency, intensity, and duration The WHO definition further stated that the aim of care in normal birth is to achieve a healthy mother and child with the least possible level of interventions, and in every case, there should be a valid reason to interfere with the natural process.

The presence of changes in cervical effacement, dilation, position, consistency, and descent of the presenting part are the key indicators in identifying the stages of labour. Concomitant with the increased frequency of contractions, a patient perceives the descent of the fetus into her pelvis as lightening (3).

The process from the 1st to the 3rd stage is a continuum without any break. The first stage of labour is the beginning and longest stage and largely determines the outcome of the labour process because commonly, a normal first stage is followed by a normal 2nd and 3rd stages of labour. Hence, in current clinical practice, the management of labour virtually equates to the management of the first stage. The pain associated with labour is a unique and complex phenomenon. Whilst typical experiences of pain tend to be associated with injury or disease, labour pain emerges during a vital and highly positive event. In fact, as the pain intensity rises, the labour is seen to be progressing normally.

The clinical audit is the systematic and critical analysis of the quality of medical care, including the procedures used for diagnosis and treatment, the use of resources and the resulting outcome and quality of life for the patient.

Reviewing of care included three domains "structure, process and outcomes" which are selected and evaluated in a systematic way according to explicit criteria .

This definition highlights two key features of the process of audit. First, audit involves a criticism of current practice. Second audit is not restricted to the technical accuracy of diagnosis or treatment but also involves diverse issues such as for example the timeliness of interventions, the appropriateness of referral, the attitudes of staff or the information given to the patient the aim of the study To improve service and quality for patients of the normal labour in the department of Obstetrics and Gynecology, Dakhla Hospital.

To assess and evaluate the practices, procedures, and outcomes of normal labor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with full-term labour that included all women who will be fullfilling the following criteria:

  * Age from 18 -40 years,
  * gestational age: complete 37 weeks gestation-41ws+6 days,
  * True labour pain associated with cervical changes, Cervical dilation > 3 cm

Exclusion Criteria:

* Multiple gestations, Fetal malformations, Complicated pregnancy (hypertension, diabetes. etc...), Intrauterine growth restriction or macrosomic fetuses, Antepartum hemorrhage or presence of meconium-stained fluid, Preterm labour and false labour pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with full-term labour that included all women who will be fullfilling the following criteria:
  * Age from 18 -40 years,
  * gestational age: complete 37 weeks gestation-41ws+6 days,
  * True labour pain associated with cervical changes, Cervical dilation > 3 cm
Sampling Method: Probability Sample
Enrollment: 176 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Maternal outcomes | 7 days
  post-partum hemorrhage percentage